CLINICAL TRIAL: NCT03698578
Title: Correlation Between Creatine Kinase Levels and Clinical and Functional Parameters in the Moments Following the Fight in Parajiu-jitsu Athletes: A Controlled Clinical Trial
Brief Title: Creatine Kinase Levels and Clinical and Functional Parameters in Parajiu-jitsu Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Jaqueline Santos Silva, Principal Investigator, São Paulo State University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: SaoPSU_UFMT1
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Healthy; Deficiency Diseases
MeSH Terms: conditions — Deficiency Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 combat fight (Experimental): Consisting of professional, high-performance paratletas. Intervention: Jiu-jitsu heating with light intensity was used for 5 minutes. The simulated fight protocol occurred in accordance with the rules of the Brazilian Confederation of Sports Jiu-Jitsu, excluding any types of finalization. In these cases, the athletes were separated and oriented to return immediately. Thus, maximum effort was advocated as well as, similar time of activity for all
  Interventions: Other: combat fight
- group 2 combat fight (Experimental): Constituted by amateur paratroopers. Intervention: Jiu-jitsu heating with light intensity was used for 5 minutes. The simulated fight protocol occurred in accordance with the rules of the Brazilian Confederation of Sports Jiu-Jitsu, excluding any types of finalization. In these cases, the athletes were separated and oriented to return immediately. Thus, maximum effort was advocated as well as, similar time of activity for all
  Interventions: Other: combat fight

INTERVENTIONS:
Other: combat fight — Jiu-jitsu heating with light intensity was used for 5 minutes. The simulated fight protocol occurred in accordance with the rules of the Brazilian Confederation of Sports Jiu-Jitsu, excluding any types of finalization. In these cases, the athletes were separated and oriented to return immediately. Thus, maximum effort was advocated as well as, similar time of activity for all

SUMMARY:
Introduction: Evidence indicates that muscle damage caused by exercise can lead to functional, biochemical and clinical damage. Therefore, it is pertinent to perform investigations related to the muscle damage marker, creatine kinase with clinical and functional responses. These outcomes encompass an intrinsic potential for understanding the real magnitude of interpretation of classic signals in athletic environments and monitoring of athletes, contributing to specific actions. Objective: To verify the correlation between clinical signs (pain and perception of recovery), functional (muscular strength) and the behavior of CK levels, in the moments following a simulated fight. METHODS: Six male parajiu-jitsu practitioners (34-44 years) were included in the study. The participants attended the collection site 4 times, with a 24-hour interval between sessions, characterizing the following collection moments: baseline, post-exertion, 24, 48 and 72 hours after the simulated fight. Data on pain (visual analogue scale - EVA), perception of recovery (Likert Scale), muscle strength (Dynamometry) and blood samples for CK analysis were collected. All parameters described were measured at all times of collection. For the analysis of the association between behavior of CK levels, clinical and functional variables, the Odds Ratio test and 95% confidence interval were used. For the gross values, the Pearson test was used according to the normality of the data.

DETAILED DESCRIPTION:
Participants will be intentionally allocated into two groups, G1 consisting of professional athletes and G2 consisting of amateur athletes. This division was carried out to guarantee homogeneous stratification between participants with level of conditioning and similar training. The anonymity of the participants will be guaranteed. There will be masking of the participants, investigator and evaluator of the results that were blind to the hypotheses and allocation in groups, adopted in the study. All participants regularly attended the same training center and no sports injuries that might compromise athletic performance will be reported during the survey.

ELIGIBILITY:
Inclusion Criteria:

* Jiu-Jitsu paratroopers were included. To be included in the study participants should report absence of anemia, inflammation, diabetes, cardiovascular disease, and musculoskeletal injuries in the six months prior to data collection. In addition, participants were instructed to refrain from anti-inflammatory drugs, analgesics, alcoholic beverages, and tobacco and did not perform any extra exercise during the study.

Exclusion Criteria:

* withdrawal of participants for personal reasons

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-02-20 (Estimated); Study Completion 2019-03-20 (Estimated)

PRIMARY OUTCOMES:
creatine kinase | post fight - 72 hours
  blood collection

SECONDARY OUTCOMES:
perception of recovery | post fight - 72 hours
  scale
muscle pain | post fight - 72 hours
  scale

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Michelletti, master, Study Chair — Paulista State University
Locations (1):
- Rayana Loch Gomes, Barra do Garças, Mount, Brazil

IPD SHARING:
Plan to Share IPD: No